CLINICAL TRIAL: NCT02953002
Title: The Correlation Between The New Sepsis Scores - SOFA, Quick SOFA and Calibrated Automated Thrombogram Values
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Elias mazen, professor, HaEmek Medical Center, Israel
Other Study IDs: EMC131-16
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Sepsis; Coagulopathy
MeSH Terms: conditions — Sepsis; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Calibrated Automated Thrombogram (CAT) — The Calibrated Automated Thrombogram (CAT). Thrombogram describes the concentration of thrombin in clotting plasma and is therefore a general physiologic function test of the thrombotic hemostatic system. The CAT measures thrombotic as well as bleeding tendency.

SUMMARY:
In total 200 subjects with diagnosis of sepsis, are planned for inclusion in this trial. After signing an informed consent a blood sample will be obtained from each participant. The investigators will measure the thrombin generation in plasma assessed by the calibrated automated thrombogram (CAT). Sequential Organ Failure Assessment score SOFA will be calculated. The relation between SOFA score and thrombin measurements will be determined.

ELIGIBILITY:
Inclusion Criteria:

* age above 18
* sepsis diagnosis

Exclusion Criteria:

* oncology patient.
* anticoagulant treatment
* pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 men and womens diagnosed with sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01-17 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
correlation between sofa score and thrombin generation | one week

CONTACTS AND LOCATIONS:
Locations (1):
- Emek medical center, Afula, Israel